CLINICAL TRIAL: NCT03011866
Title: Intravenous Versus Topical Use of Tranexamic Acid in Reducing Gross Hemorrhage and Transfusions of Spine Surgeries (TARGETS) : A Prospective, Randomized, Double Blind, Head-to-head Comparison Study
Brief Title: Tranexamic Acid in Reducing Gross Hemorrhage and Transfusions of Spine Surgeries
Acronym: TARGETS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Shugang Li, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PUMCH-000391
Record Dates: First submitted 2016-12-16; First posted 2017-01-05 (Estimated); Last update posted 2017-01-05 (Estimated); Status verified 2017-01

CONDITIONS: Spinal Stenosis; Intervertebral Disc Displacement
MeSH Terms: conditions — Spinal Stenosis; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental (Experimental): Loading dose: 100ml 0.9% normal saline(NS) intravenous infusion, 15-20min prior to operation initiation.
  Maintenance dose: 5ml/hr 0.9% NS intravenous infusion till the last suture. Bolus dose: the wound topically irrigated with 500mg TXA in 250ml 0.9% NS for 5min. Waste fluid was then removed by suction, and the wound was closed.
  Interventions: Drug: Wound topically irrigated with 500mg TXA
- Control (Other): Loading dose: 10mg/kg tranexamic acid(TXA) in 100ml 0.9% NS intravenous infusion, 15-20min prior to operation initiation.
  Maintenance dose: 1mg/kg/hr TXA intravenous infusion till the last suture. Bolus dose: the wound topically irrigated with 250ml 0.9% NS for 5min. Waste fluid was then removed by suction, and the wound was closed.
  Interventions: Drug: 1mg/kg/hr TXA intravenous infusion till the last suture

INTERVENTIONS:
Drug: Wound topically irrigated with 500mg TXA
  Arms: Experimental
Drug: 1mg/kg/hr TXA intravenous infusion till the last suture
  Arms: Control

SUMMARY:
Multilevel decompression and bone graft fusion is a most effective measure for treating degenerative lumbar spinal diseases. Yet, the surgery is commonly associated with large amount of perioperative blood loss and high demand for homologous blood transfusion. Tranexamic acid (TXA) has been proved as efficient in reducing the gross blood loss in various kinds of surgeries. However, high quality evidence of its efficacy and safety is still lacking in lumbar spinal surgeries. Besides, systemic use of TXA carries the risks of thromboembolic complications such as deep venous thrombosis and pulmonary embolism, thus the optimal drug delivery route of TXA remains undetermined. The aim of this study is to test the non-inferiority of topical TXA application to its intravenous use in multilevel decompression and bone graft fusion surgeries. A prospective, randomized, double-blind, head-to-head comparison study design will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists(ASA)classification of physical status I-II.
* Aged over 50yrs.
* Patients suffering from spinal stenosis or intervertebral disc displacement and require multilevel decompression and bone graft fusion surgeries.
* Written informed consent.

Exclusion Criteria:

* ASA III-IV.
* Age≤ 50yrs.
* History of chronic renal dysfunction (preoperative blood creatinine> 120mmol/L), liver dysfunction (preoperative blood aspartate or alanine aminotransferase> 50 units/L) or history of coronary artery disease with stent placement.
* Abnormal preoperative coagulation profile (preoperative prothrombin time elongation> 3s, activated partial thromboplastin time elongation> 10s, platelet counts< 100*10^9/L or >400*10^9/L, or INR> 1.4).
* Pre-existing anemia (male< 12g/dL, female<11g/dL).
* Long-term medications of aspirin and/or other anticoagulants.
* Patients known as allergic to TXA.
* Patients who have religious and/or other beliefs limiting blood transfusion.
* Dura mater laceration and/or unexpected massive bleeding during operation.
* Cell saver application during operation.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2017-02; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Perioperative Total blood loss (TBL) | Since operation initiation till postoperative day 3 (POD3)
  TBL= PBV*（hematocrit on postoperative day 3- preoperative hematocrit）/average hematocrit; Predicted blood volume(PBV)= k1* height^3(m)+ k2* weight(kg)+ k3 (female: k1=0.3561， k2=0.03308， k3=0.1833, male: k1=0.3669， k2=0.03219， k3=0.6041)

SECONDARY OUTCOMES:
Visible intraoperative blood loss | Since operation initiation till operation completion, an average of 120min
Visible postoperative blood loss within 24hrs | 0- 24hrs postoperatively
Visible postoperative blood loss within 48hrs | 0- 48hrs postoperatively
Combined visible perioperative blood loss | Since operation initiation till postoperative 48hrs
  Combined visible perioperative blood loss= visible intraoperative blood loss + visible postoperative blood loss within 24hrs + visible postoperative blood loss within 48hrs
Total postoperative blood loss | 0- 48hrs postoperatively
  Total postoperative blood loss= drainage day1(ml)* drainage Hct day1(%)/blood Hct day1(%)+ drainage day2(ml)* drainage Hct day2(%)/blood Hct day2(%)
Postoperative hidden blood loss (HBL) | 48hrs postoperatively
  HBL=TBL- combined visible perioperative blood loss
Postoperative prothrombin time(PT) | Tested at operation completion, postoperative 24hrs and postoperative 48hrs
Postoperative activated partial thromboplastin time(APTT) | Tested at operation completion, postoperative 24hrs and postoperative 48hrs
Postoperative fibrinogen level(Fbg) | Tested at operation completion, postoperative 24hrs and postoperative 48hrs
Postoperative international normalized ratio(INR) | Tested at operation completion, postoperative 24hrs and postoperative 48hrs
Postoperative R time | Tested at operation completion, postoperative 24hrs and postoperative 48hrs, using thromboelastography tests.
Postoperative K time | Tested at operation completion, postoperative 24hrs and postoperative 48hrs, using thromboelastography tests.
Postoperative maximum amplitude (MA) | Tested at operation completion, postoperative 24hrs and postoperative 48hrs, using thromboelastography tests.
Postoperative lysis after 30 minutes(LY 30) | Tested at operation completion, postoperative 24hrs and postoperative 48hrs, using thromboelastography tests.
Postoperative hemoglobin nadir | Since operation completion till postoperative 48hrs
Perioperative transfusion rates | Since operation initiation till postoperative 48hrs
Perioperative transfusion amounts | Since operation initiation till postoperative 48hrs
Length of hospital stay | A single inpatient duration since the day of admission till the day of discharge, an average of 1 week
  Length of hospital stay is calculated by subtracting day of admission from day of discharge.
Adverse event rates | Since operation initiation till postoperative 48hrs
  Adverse events include deep venous thrombosis, myocardial infarction, pulmonary embolism, cerebrovascular disease, impaired liver function, impaired renal function and incisional hematoma/ infection.

REFERENCES:
- [Derived] Hui S, Tao L, Mahmood F, Xu D, Ren Z, Chen X, Sheng L, Zhuang Q, Li S, Huang Y. Tranexamic Acid in Reducing Gross Hemorrhage and Transfusions of Spine Surgeries (TARGETS): study protocol for a prospective, randomized, double-blind, non-inferiority trial. Trials. 2019 Feb 12;20(1):125. doi: 10.1186/s13063-019-3231-9. PMID 30755256